CLINICAL TRIAL: NCT00706680
Title: The Use of Thymoglobulin in a Calcineurin Inhibitor and Steroid Minimization Protocol
Brief Title: Thymoglobulin in Calcineurin Inhibitor and Steroid Minimization Protocol
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Genzyme, a Sanofi Company (Industry); Unity Health Toronto (Other); St. Paul's Hospital, Canada (Other)
Responsible Party: Dr. Edward Cole, University Health Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 07-0619-A
Record Dates: First submitted 2008-02-08; First posted 2008-06-27 (Estimated); Last update posted 2008-06-27 (Estimated); Status verified 2008-02

CONDITIONS: Diabetes; Graft Rejection
MeSH Terms: conditions — Diabetes Mellitus | interventions — thymoglobulin; Methylprednisolone Hemisuccinate; Steroids; Prednisone; Mycophenolic Acid; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): All subjects meeting the entry criteria will be treated with the study immunosuppressive protocol.
  Interventions: Drug: Thymoglobulin

INTERVENTIONS:
Drug: Thymoglobulin — methyl prednisone intravenously pre-operatively, as per institutional practice. Thymoglobulin, initiated prior to completion of the anastomosis, or if not possible, within 24 hours of transplantation for a total dose of 6-7.5mg/kg given over 3-5 doses. Steroids initiated post-operatively at 1mg/kg/day for 2 days, then 0.5mg/kg/day for 2 days, then 0.25mg/kg/day for 2 days. Patients will be placed on 5mg daily for the remainder of the study. All patients will receive Mycophenolic acid at a dose of 2gm/day (Cellcept) or 1440mg/day (Myfortic) post-transplantation with dose adjustment as needed. Cyclosporine micro-emulsion will be initiated when renal function is established or no later than day 10 in a dose of 3mg/kg twice daily with adjustment to achieve a C2 target of 600-800 nanograms/ml.
  Other Names: Thymo; Polyclonal ATG; Methyl Prednisone; SoluMedrol; Steroid; Prednisone; MMF; Cell Cept; Mycophenolate Mofetil; Mycopnlolic Acid; Myfortic; Cyclosporine; Neoral

SUMMARY:
This study has been designed to test whether using Thymoglobulin with low dose Cyclosporine and early steroid dosage reduction will minimize both kidney rejection and the development of new onset diabetes mellitus after renal transplant.

DETAILED DESCRIPTION:
All patients will receive methyl prednisone intravenously pre-operatively, as per institutional practice. Thymoglobulin will be initiated prior to completion of the anastomosis, or if not possible, within 24 hours of transplantation in all patients and a total dose of 6-7.5mg/kg will be given over 3-5 doses. Steroids will be initiated post-operatively at 1mg/kg/day for 2 days, then 0.5mg/kg/day for 2 days, then 0.25mg/kg/day for 2 days and then patients will be placed on 5mg daily for the remainder of the study. All patients will receive Mycophenolic acid at a dose of 2gm/day (Cellcept) or 1440mg/day (Myfortic) post-transplantation with dose adjustment as needed. Cyclosporine micro-emulsion will be initiated when renal function is established or no later than day 10 in a dose of 3mg/kg twice daily with adjustment to achieve a C2 target of 600-800 nanograms/ml.

ELIGIBILITY:
Inclusion Criteria:

* De Novo, single Kidney recipient
* At least 1 HLA mismatch

Exclusion Criteria:

* Recipient of multiple organs
* prior transplant recipient
* Subjects who have Diabetes prior to transplant, as indicated by pre-transplant OGTT
* PRA >10%
* Hepatitis B surface antigen positive
* Hepatitis C antibody positive
* HIV positive

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-02 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients developing New Onset Diabetes post transplant, as identified by an oral glucose tolerance test | 6 months post transplant.

SECONDARY OUTCOMES:
Incidence of acute rejection | 6 months post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Edward Cole, Study Director — University Health Network, Toronto; John Gill, Principal Investigator — St. Paul's Hospital; Ramesh Prasad, Principal Investigator — Unity Health Toronto
Locations (3):
- Canada (3):
  - St Paul's Hospital, Vancouver, British Columbia
  - St Michael's Hospital, Toronto, Ontario
  - University health Network, Toronto, Ontario

REFERENCES:
- [Derived] Cole EH, Prasad GV, Cardella CJ, Kim JS, Tinckam KJ, Cattran DC, Schiff JR, Landsberg DN, Zaltzman JS, Gill JS. A pilot study of reduced dose cyclosporine and corticosteroids to reduce new onset diabetes mellitus and acute rejection in kidney transplant recipients. Transplant Res. 2013 Jan 12;2(1):1. doi: 10.1186/2047-1440-2-1. PMID 23369458